CLINICAL TRIAL: NCT06549075
Title: Efficacy of a Personalized Modular Intervention to Promote Dignity, Meaningfulness and Mindfulness by a Palliative Care Consultation-Liaison Service in Swiss Acute Hospital Care. A Randomized Controlled Trial
Brief Title: Therapeutic Support to Strengthen Dignity, Mental Well-being and Quality of Life in Acute Palliative Care Patients.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-01301; 2024-01301 (Other: Ethics Committee North and Central Switzerland)
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Promoting Dignity, Meaningfulness and Mindfulness in Acute Palliative Care
MeSH Terms: interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personnalized modular therapeutic support (Experimental)
  Interventions: Other: Therapeutic support; Other: Standard Specialized Palliative Consultation Service
- Standard Specialized Palliative Consultation Service (Active Comparator)
  Interventions: Other: Standard Specialized Palliative Consultation Service

INTERVENTIONS:
Other: Therapeutic support — The modular intervention consists of three modules, including Dignity Therapy, CALM Therapy and Mindfulness-based training. According to the patient's preferences, the patient will be allocated to one of the three interventions, which will be conducted by trained therapists within two sessions.
  Other Names: personnalized modular therapeutic support
  Arms: Personnalized modular therapeutic support
Other: Standard Specialized Palliative Consultation Service — According to needs standard specialized palliative care will include support of symptom control, shared decision making/ advance care planning, network planning and support of relatives.

SUMMARY:
The goal of this clinical trial is to test the benefit of a newly designed personalized therapeutic intervention compared to the standard specialized palliative care service at the swiss acute palliative hospital care.The main questions it aims to answer are:

Does an additional therapeutic support that fits the individual needs of a palliative care patient increases dignity and mental well-being as measures by a questionnaire (Patient Dignity Inventory) to a larger extent than standard palliative care alone? Is the additional therapeutic support perceived as helpful? Researchers will compare the additional therapeutic support with standard palliative care to standard palliative care alone.

Participants will:

Receive additional therapeutic support in two structured sessions a 60 minutes and/or standard palliative care Fill out questionnaires before and after therapeutic interventions and standard palliative care Provide a semi-structured interview following the therapeutic support

DETAILED DESCRIPTION:
Patient with a life-limiting serious illness commonly experience substantial emotional and spiritual distress, death anxieties, depressive symptoms and loss of dignity and purpose in life. Fostering dignity and meaning and relieving psychological distress have been identified as a core objective for end-of-life care. However, individual's needs for dignity and psychological support at the end of life may vary. Therefore, a personalized approach is needed. On the basis of theoretical frameworks and existing dignityfostering and meaning based interventions, and a workshop with international experts in the field of palliative care, we have developed a personalized modular intervention, consisting of three modules, including CALM Therapy, Dignity Therapy, and a mindfulness-based intervention.

The overall purpose of this study is to test the efficacy of the designed personalized modular intervention compared to the specialized palliative care service at the swiss acute palliative hospital care.

Patients are randomized to either receiving standard specialized palliative consultation (SSPC) and the modular intervention or standard palliative consultation services alone. Within the intervention group, participants can choose one of the three modules based on personal preference and the recommendation of the palliative care team (based on assessment). All three interventions consist of two structured sessions.

The control group will receive SSPC alone. According to needs standard specialized palliative care will include support of symptom control, shared decision making/ advance care planning, network planning and support of relatives.

SSPC is performed by specialized inter-professional palliative care service, including doctors and advanced nurse practitioners, certified by national standards for specialist palliative care. Other professions are involved depending on needs. Patients are seen as required at least twice a week.

Patients will be asked to fill in a set of questionnaires at baseline (T0), after the completion of the intervention (T1) and at 1-month follow-up (T2). A brief semi-structured qualitative interview will be conducted with the patients following completion of the intervention to assess perceived benefits and challenges of the intervention.

The primary objective is to evaluate if mental well-being tend to improve over the pre- versus post study design as measured by the Patient Dignity Inventory and if this effect is significantly larger in the modular intervention group as compared to the standard specialized palliative consultation (SSPC) group.

ELIGIBILITY:
Inclusion criteria:

* Informed Consent
* Patients seen by the palliative consultation-liaison service at the University Hospital Basel as an in- or outpatient
* Suffering from a life-limiting serious illness (≤ 18 months)
* ≥ 18 years of age
* Willingness and capacity to commit to three study visits

Exclusion criteria:

* Delirious (ICD-10: F05.9)
* Inability to give consent (lack of decisional capacity to consent)
* Inability to follow the procedures of the study due to psychological disorders, dementia, or other cognitively impairment of the participant,
* Too ill to complete the requirements of the protocol
* Unable to understand, speak and read German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient Dignity Inventory | Baseline, after intervention, 4 week follow-up
  Questionnaire (Self-reported outcome)